CLINICAL TRIAL: NCT03124498
Title: A Phase I/II, Open Label Study to Evaluate the Safety and Efficacy of Autologous Cytokine-Induced Killer (CIK) Cell for Patients With Hepatocellular Carcinoma (HCC) After Transarterial Chemoembolization (TACE), Percutaneous Ethanol Injection Therapy (PEIT) or RadioFrequency Ablation (RFA) Therapy
Brief Title: A Study to Evaluate Autologous CIK Cells in Patients With Hepatocellular Carcinoma After TACE, PEIT or RFA
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chuan An Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CABIO-CIK-1701
Record Dates: First submitted 2017-04-19; First posted 2017-04-21 (Actual); Last update posted 2017-04-21 (Actual); Status verified 2017-04

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma, Autologous Cytokine-Induced Killer
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CIK Cell (Experimental): Phase I - Three dose levels escalated according to 3+3 rule
  Phase II - The recommended dose level according to the results from Phase I
  Interventions: Biological: CIK Cell

INTERVENTIONS:
Biological: CIK Cell — Autologous cytokine-induced killer (CIK) cell

SUMMARY:
A Phase I/II, Open Label Study to Evaluate the Safety and Efficacy of Autologous Cytokine-Induced Killer (CIK) Cell for Patients with Hepatocellular Carcinoma (HCC) after Transarterial Chemoembolization (TACE), Percutaneous Ethanol Injection Therapy (PEIT) or RadioFrequency Ablation (RFA) Therapy.

ELIGIBILITY:
Inclusion Criteria:

1. 20 to 80 years old men and women;
2. HCC diagnosed with typical imaging findings, or confirmed by needle liver biopsy;
3. Patients who are not a transplant candidate;
4. Patients who have no extrahepatic metastasis and are with measurable residual tumor after TACE, PEIT or RFA therapy;
5. Patients who have a life expectancy of at least 6 months;
6. Child-Pugh Class should be A or B;
7. Eastern Cooperative Oncology Group (ECOG) performance status score was 0-3;
8. Patients who have clinical laboratory test results as follows:

   * Absolute neutrophil count ≥ 1,500/µL or White blood cell ≥ 4,000/µL
   * Hemoglobin ≥ 8.5 g/dL
   * Platelet count ≥ 50,000/µL
   * Blood creatinine ≤ 1.5 x upper limit of normal
   * Total bilirubin < 3 x upper limit of normal
   * Albumin ≥ 2.8 g/dL
   * International normalized ratio (INR) / Partial thromboplastin time (PTT) < 1.5 x upper limit of normal
9. Written informed consent.

Exclusion Criteria:

1. Patients who have infiltrative or diffuse HCC;
2. Patients who have significant cardiovascular disease such as myocardial infarction occurred within recent 6 months, chronic heart failure or unstable coronary artery disease;
3. Patients who plan to receive systemic chemotherapy or target therapy;
4. Patients with other malignant tumor within the past 5 years before treatment;
5. Pregnant or lactating patients;
6. Patients with hemorrhage/bleeding event;
7. Patients with uncontrolled infections;
8. Known or suspected allergy to the investigational agent or any agent given in association with this trial;
9. Patients who have current Human Immunodeficiency Virus (HIV) or Treponema Pallidum (TP) infection;
10. Patients who are suffering from serious autoimmune disease;
11. Patients who have had long term use of or are using an immunosuppressant;
12. History of organ transplant;
13. Prior use of any anti-cancer treatments within 30 days or 5 half-lives (whichever is longer), except TACE, PEIT and RFA therapy;
14. Patients who have participated in another clinical study and received treatment within 30 days prior to the screening visit;
15. Mental conditions rendering the patient incapable of understanding the nature, scope, and consequences of the study;
16. Other situations that the researchers considered unsuitable for this study.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2017-11 (Estimated); Primary Completion 2019-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Phase I: Presence or absence of Dose-Limiting Toxicity | 5 Weeks
Phase II: Disease Control Rate | 24 Weeks